CLINICAL TRIAL: NCT02034786
Title: Phase I Study of a Filler Agent Composed of Mesenchymal Stem Cells Obtained From Autologous Adipose Tissue Associated With Hyaluronic Acid
Brief Title: Safety Study of Filler Agent Composed of Autologous Mesenchymal Stem Cells and Hyaluronic Acid
Acronym: LipAge
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cryopraxis Criobiologia Ltda. (Industry)
Collaborators: Hospital Federal de Bonsucesso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cryo 394.191; 394.191 (Other: CEP)
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Lipodystrophies; Aesthetics Procedure
Keywords: Mesenchymal stem cell; Hyaluronic acid; Adipose Tissue; Filler Agent
MeSH Terms: conditions — Lipodystrophy | interventions — Administration, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Adipose tissue collection and Transdermal injection of the filler agent, composed of mesenchymal stem cells derived from the autologous adipose tissue, associated with hyaluronic acid.
  Interventions: Procedure: Adipose tissue collection; Biological: Transdermal injection
- Control (Active Comparator): Transdermal injection of hyaluronic acid only.
  Interventions: Procedure: Transdermal injection

INTERVENTIONS:
Procedure: Adipose tissue collection — Only the patients selected for the Test Group will go through the procedure. The adipose tissue collection will occur in an elective surgery liposuction, in patients who meet the inclusion criteria, after signing the informed consent form. Thus, the material that would be disposed after surgery will be donated to the study.
  The material for the study will be collected by the tumescent liposuction technique, which involves the removal of subcutaneous fat under local anesthesia.
  Arms: Test
Biological: Transdermal injection — Transdermal injection of the filler agent composed of mesenchymal stem cells derived from autologous adipose tissue associated with hyaluronic acid.
  Arms: Test
Procedure: Transdermal injection — Transdermal injection of hyaluronic acid only.
  Arms: Control

SUMMARY:
Lipodystrophies are part of a clinically heterogeneous group of disorders characterized by loss (lipoatrophies) and / or accumulation of fat, which usually results in a change of normal tissue surface. Millions of plastic and reconstructive surgeries are performed annually to repair soft tissue defects due to trauma, tumor resection and congenital defects. Surgical options for lipoatrophy, the lipodystrophy type characterized by subcutaneous adipose tissue atrophy, include: Transfer of autologous fat, Dermis - fat graft, Skin flaps and Commercially available fillers.

Currently, the most commonly filler agent used for the lipodystrophy treatment is polymethylmethacrylate, considered permanent and with a history of short- and medium-term adverse effects. Biocompatible and temporary filler agents such as hyaluronic acid, polylactic acid and collagen have been used for over 25 years for cosmetic purposes and in lipoatrophies. More recently, the use of autologous fibroblasts proved to be efficient solving acne scars and enabling dermis regeneration. Studies in mice showed that the combination of pre - adipocytes with a biomaterial is much more effective in tissue reconstitution than the injection of adipose tissue only, providing volume and also stimulating cell proliferation and differentiation with increased production of extracellular matrix.

This project aims a phase I clinical trial of a filler agent, composed of mesenchymal stem cells derived from autologous adipose tissue associated with hyaluronic acid.

DETAILED DESCRIPTION:
Open, controlled and randomized study. The intervention performed in this study will be the transdermal injection of the filler agent in patients undergoing elective cosmetic liposuction procedure, with legal age and without any of the exclusion criteria items. Patients will be evaluated according to the parameters for a total period of 12 months.

Individuals in the control group will have transdermal injection of hyaluronic acid and will be evaluated with the same parameters used for the study group and also for the same period.

In this study, 25 volunteers attended at Dermatologic Service of the Bonsucesso Federal Hospital (HFB) will be included.

The research subjects will be evaluated preliminarily regarding inclusion and exclusion criteria of the study and the procedure will only be performed after the signing of the Informed Consent Form (ICF).

The efficacy and safety study will be conducted following Good Laboratory and Clinics Practices.

Patients who meet the study eligibility criteria will be randomly assigned to one of the two treatment groups: Test or Control.

The first follow-up visit will occur in the first month post-procedure. Subsequent consultations will be held at 3, 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years;
* Signature of the ICF;
* Suitable for the following preoperative laboratory tests results: complete blood count, coagulation, biochemistry, electrocardiogram, hepatogram and β-human chorionic gonadotropin (hCG) for women of childbearing age.

Exclusion Criteria:

* Patients unable to undergo surgery liposuction with Klein technique as those with severe cardiovascular disease, severe coagulation disorders including thrombophilia and pregnancy;
* Patients with limited understanding of the procedure;
* Pregnant or lactating;
* Under 18 years;
* Immunosuppressed;
* Lack of signature of the ICF;
* Use of drugs;
* Patients with preoperative results considered inadequate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events Analysis | Every visit over the first 12 months after intervention
  Proportion of patients with non-serious and serious adverse events in the first 12 months after the intervention.

SECONDARY OUTCOMES:
Efficacy Analysis | 1, 3, 6 and 12 months after the intervention
  Difference of volume increase, captured by images, between control and study group at different times after the intervention (1, 3, 6 and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RC Souza, M.D, Principal Investigator — Dermatology Service
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro, Brazil